CLINICAL TRIAL: NCT01912911
Title: Evaluating the Efficacy and Feasibility of a Novel Wireless ECG Recording System in Monitoring Patients After Atrial Fibrillation Ablation Procedure
Acronym: iTransmit
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Khaldoun Tarakji, MD MPH, The Cleveland Clinic
Other Study IDs: 13-521
Record Dates: First submitted 2013-06-07; First posted 2013-07-31 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Persistent Atrial Fibrillation; Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators goal in this study is to examine the feasibility and efficacy of AliveCor iphone case monitoring device in monitoring patients after AF ablation by comparing transmissions using Alive Cor with transmissions from a traditional transtelephonic monitor (TTM).

A secondary goal is to assess the ease of use of AliveCor device compared to traditional TTM system from the patient's perspective

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between > 18 and < 75 years of age
2. Paroxysmal or persistent atrial fibrillation
3. Scheduled to undergo an AF ablation procedure
4. Already has iPhone 4 or iPhone 4S with data plan
5. Willing to use the iPhone Alive Cor case
6. Written informed consent

Exclusion Criteria:

1. Unable or unwilling to use the Alive Cor case for their iPhone or iPhone 4S
2. Residing outside the United States

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing A-fib ablations.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The proportion of AF/flutter events detected by the AliveCor device will be compared to events detected by the TTM for each episode. | 3 months

SECONDARY OUTCOMES:
Amount of transmissions from smartphone in comparison with traditional TTM method | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Khaldoun Tarajki, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic HVI, Cleveland, Ohio, United States